CLINICAL TRIAL: NCT01208545
Title: Serial Electrophysiologic Monitoring During Administration of Nerve-Toxic Chemotherapeutic Drugs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NeuroMetrix, Inc. (Industry)
Responsible Party: Eugene A. Lesser, D.O., Senior Medical Director, NeuroMetrix, Inc.
Other Study IDs: 99000287
Record Dates: First submitted 2010-09-22; First posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Chemotherapy; Nerve Degeneration; Nerve Conduction
Keywords: taxol; vincristine; oxaliplatin; chemotherapy; nerve degeneration; nerve conduction; cancer; nerve conduction studies
MeSH Terms: conditions — Nerve Degeneration; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study hypothesis is that changes in serially obtained nerve conduction study data obtained every 3-4 weeks in cancer patients receiving chemotherapy can be used to predict the development of a clinically significant / disabling drug induced neuropathy six and twelve months following the start of treatment. Patients with breast cancer, colon cancer, gastroesophageal cancer, and non-Hodgkins lymphoma will be enrolled. Six lower extremity nerves--three in each leg--will be electrically stimulated and their responses recorded at three to four week intervals coinciding with patient's scheduled chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of untreated breast cancer, treated (advance stage) or untreated colon cancer, untreated non-Hodgkins lymphoma, or advanced gastroesophageal cancer scheduled to begin chemotherapy with either Taxol, oxaliplatin, or vincristine

Exclusion Criteria:

* Individuals with an implanted electronic medical devices (cardiac pacemaker or defibrillator, vagus nerve stimulator, deep brain stimulator, intrathecal pump, others)
* Individuals whose chemotherapy regimen will include nerve toxic drugs other than Taxol, oxaliplatin, or vincristine, or includes more than one of these three drugs in combination
* Individuals whose screening nerve conduction studies show peroneal motor amplitude < 1 mV bilaterally or sural sensory amplitude < 3 uV bilaterally or no result obtainable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to an oncology clinic for treatment of breast cancer, colon cancer, or non-Hodgkins lymphoma, or treatment of advanced gastroesophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Time in weeks to fifty percent decrease in sural nerve action potential amplitude | one year

CONTACTS AND LOCATIONS:
Overall Officials: Eugene A Lesser, D.O., Principal Investigator — NeuroMetrix, Inc.
Locations (1):
- Santa Clara Valley Health and Hospital System, Santa Clara, California, United States